CLINICAL TRIAL: NCT00849693
Title: A Double-Blind, Efficacy and Safety Study of Duloxetine Versus Placebo in the Treatment of Children and Adolescents With Major Depressive Disorder
Brief Title: A Study in the Treatment of Children and Adolescents With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7109; F1J-MC-HMCL (Other: Eli Lilly and Company); NCT00892294 (obsolete NCT alias)
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fluoxetine (Active Comparator)
  Interventions: Drug: fluoxetine
- Duloxetine 60 mg (Experimental)
  Interventions: Drug: duloxetine
- Duloxetine 30 mg (Experimental)
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: Placebo — Capsules identical in appearance, color, taste, and smell to study drug, orally, once daily for 10 weeks (acute treatment phase)
  Arms: Placebo
Drug: fluoxetine — 20 milligram (mg) orally, once daily for 10 weeks (acute treatment phase) and 20-40 mg orally, once daily for additional 6 months (extension phase)
  Other Names: LY110140; Prozac
  Arms: Fluoxetine
Drug: duloxetine — 60 mg orally, once daily for 10 weeks (acute treatment phase) and 60-120 mg orally, once daily for additional 6 months (extension phase)
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 60 mg
Drug: duloxetine — 30 mg orally, once daily for 10 weeks (acute treatment phase) and 60-120 mg orally, once daily for additional 6 months (extension phase)
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 30 mg

SUMMARY:
The purpose of this study is to assess whether duloxetine is superior to placebo in the treatment of children and adolescents with major depressive disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, diagnosed with major depressive disorder (MDD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and supported by the Mini International Neuropsychiatric Interview for children and adolescents (MINI-KID).
* Diagnosis of moderate or greater severity of MDD as determined by Children's Depression Rating Scale - Revised (CDRS-R) with a total score greater than or equal to 40 at screen, and randomization and a Clinical Global Impression of Severity (CGI-Severity) rating of greater than or equal to 4 at screen, and randomization.
* Female patients must test negative for pregnancy during screening.
* Judged to be reliable by the investigator to keep all appointments for clinical visits, tests, and procedures required by the protocol.
* Has a degree of understanding such that they can communicate intelligently with the investigator and study coordinator.
* Capable of swallowing study drug whole. It is anticipated the patients will need to swallow up to 6 capsules per day.
* Patients must have venous access sufficient to allow blood sampling and are compliant with blood draws as per the protocol.

Exclusion Criteria:

* Children of site personnel directly affiliated with this study and/or their immediate families.
* Children of Lilly employees or employees of the designated clinical research organization (CRO) assisting with the conduct of the study.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, or pervasive development disorder, as judged by the investigator.
* Have a history of DSM-IV-TR-defined substance abuse or dependence within the past year, excluding caffeine and nicotine.
* Have a current primary DSM-IV-TR Axis I disorder other than MDD or a current secondary DSM-IV-TR Axis I disorder that requires any pharmacologic treatment
* Have 1 or more first-degree relatives with diagnosed bipolar I disorder.
* Have a significant suicide attempt within 1 year of screening or are currently at risk of suicide in the opinion of the investigator.
* Have a weight less than 20 kilogram (kg) at screening.
* Have a lack of response to 2 or more adequate treatment trials of antidepressants at a clinically appropriate dose for a minimum of 4 weeks for the same MDD episode.
* Have initiated, stopped, or changed the type or intensity of psychotherapy within 6 weeks prior to screening.
* Have a history of seizure disorder (other than febrile seizures).
* Have a history of electroconvulsive therapy within 1 year of screening.
* Have had treatment with a monoamine oxidase inhibitor (MAOI) within 14 days or fluoxetine within 30 days of randomization; or the potential need to use an MAOI during the study or within 5 weeks of discontinuation of study drug.
* Have previously enrolled, completed, or withdrawn from this study or any other study investigating duloxetine or fluoxetine.
* Have a positive urine drug screen for any substances of abuse or excluded medication.
* Are taking any excluded medications that cannot be discontinued by screening.
* Have known hypersensitivity to duloxetine, fluoxetine, or their inactive ingredients; or have frequent or severe allergic reactions to multiple medications.
* Have uncontrolled narrow-angle glaucoma.
* Have acute liver injury or severe cirrhosis.
* Have a serious or unstable medical illness, psychological condition, or clinically significant laboratory or electrocardiogram (ECG) result that, in the opinion of the investigator, would compromise participation in the study or be likely to lead to hospitalization.
* Have abnormal thyroid-stimulating hormone concentration.
* Have initiated or discontinued hormone therapy within the previous 3 months.
* Female patients who are either pregnant, nursing or have recently given birth.
* Need to use thioridazine during the study or within 5 weeks after discontinuation of study drug or need to use pimozide during the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 463 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (44):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dothan, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carson, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Imperial, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middletown, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton Twp, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salem, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dalllas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wharton, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Allis, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parry Sound, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
- Mexico (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalnepantla

REFERENCES:
- [Derived] Emslie GJ, Wells TG, Prakash A, Zhang Q, Pangallo BA, Bangs ME, March JS. Acute and longer-term safety results from a pooled analysis of duloxetine studies for the treatment of children and adolescents with major depressive disorder. J Child Adolesc Psychopharmacol. 2015 May;25(4):293-305. doi: 10.1089/cap.2014.0076. PMID 25978741
- [Derived] Emslie GJ, Prakash A, Zhang Q, Pangallo BA, Bangs ME, March JS. A double-blind efficacy and safety study of duloxetine fixed doses in children and adolescents with major depressive disorder. J Child Adolesc Psychopharmacol. 2014 May;24(4):170-9. doi: 10.1089/cap.2013.0096. Epub 2014 May 9. PMID 24815533

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 10-week acute treatment phase, and a 6-month extension phase.
Groups:
- Duloxetine 60 mg / Duloxetine 60-120 mg: Participants were treated with Duloxetine 60 milligram (mg) orally, once daily for 10 weeks during acute treatment phase and Duloxetine 60-120 mg orally, once daily for 6 months during extension phase
- Duloxetine 30 mg/Duloxetine 60-120 mg: Participants were treated with Duloxetine 30 mg orally, once daily for 10 weeks during acute treatment phase and Duloxetine 60-120 mg orally, once daily for 6 months during extension phase
- Fluoxetine 20 mg/Fluoxetine 20-40 mg: Participants were treated with Fluoxetine 20 mg orally, once daily for 10 weeks during acute treatment phase and Fluoxetine 20-40 mg orally, once daily for 6 months during extension phase
- Placebo/Duloxetine 60-120 mg: Participants were treated with placebo orally, once daily for 10 weeks during acute treatment phase and Duloxetine 60-120 mg orally, once daily for 6 months during extension phase
Period: Acute Treatment Phase
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Started | 108 | 116 | 117 | 122
Completed | 75 (2 didn't enter extension phase.) | 81 (1 didn't enter extension phase) | 84 | 85 (3 didn't enter extension phase)
Not Completed | 33 | 35 | 33 | 37
Not completed — Adverse Event | 12 | 7 | 6 | 4
Not completed — Lost to Follow-up | 5 | 8 | 11 | 9
Not completed — Protocol Violation | 1 | 5 | 2 | 6
Not completed — Withdrawal by Subject | 5 | 5 | 3 | 8
Not completed — Parent or caregiver decision | 7 | 6 | 7 | 7
Not completed — Physician Decision | 2 | 1 | 2 | 1
Not completed — Sponsor decision | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 3 | 1 | 2
Period: Extension Phase
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Started | 73 | 80 | 84 | 82
Completed | 43 | 50 | 49 | 44
Not Completed | 30 | 30 | 35 | 38
Not completed — Adverse Event | 4 | 6 | 3 | 7
Not completed — Lost to Follow-up | 7 | 5 | 6 | 6
Not completed — Protocol Violation | 0 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 6 | 9 | 10 | 15
Not completed — Parent or caregiver decision | 9 | 4 | 10 | 5
Not completed — Physician Decision | 1 | 1 | 2 | 0
Not completed — Sponsor decision | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg | Total
Number analyzed (Participants) | 108 | 116 | 117 | 122 | 463
Age Continuous [Mean (Standard Deviation); unit: years] | 12.92 (2.925) | 12.86 (2.904) | 13.04 (3.205) | 13.09 (2.895) | 12.98 (2.977)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 47 | 61 | 69 | 237
  Male | 48 | 69 | 56 | 53 | 226
Race/Ethnicity, Customized [Number; unit: Participant]
  American Indian or Alaska Native | 15 | 23 | 16 | 19 | 73
  Asian | 0 | 1 | 1 | 1 | 3
  Black or African American | 27 | 21 | 21 | 24 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White | 54 | 61 | 67 | 62 | 244
  Multiracial | 6 | 6 | 9 | 13 | 34
  Not Provided | 6 | 3 | 3 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 87 | 86 | 93 | 98 | 364
  Mexico | 16 | 25 | 16 | 17 | 74
  Canada | 5 | 5 | 7 | 7 | 24
  Argentina | 0 | 0 | 1 | 0 | 1
Children's Depression Rating Scale-Revised (CDRS-R) Total Score [Mean (Standard Deviation); unit: units on a scale] — CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression.
  units on a scale | 59.3 (10.87) | 59.8 (11.00) | 57.9 (10.11) | 58.2 (9.35) | 58.8 (10.33)
CDRS-R Subscale Scores [Mean (Standard Deviation); unit: units on a scale] — CDRS-R Subscale score include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21.
  units on a scale
    Mood | 16.6 (3.69) | 16.4 (3.64) | 16.0 (3.52) | 16.0 (3.38) | 16.2 (3.55)
    Somatic | 19.6 (4.58) | 19.7 (4.87) | 19.3 (4.60) | 19.5 (4.28) | 19.5 (4.57)
    Subjective | 10.1 (3.51) | 10.6 (3.60) | 10.0 (3.35) | 10.0 (2.79) | 10.2 (3.32)
    Behavior | 13.0 (3.04) | 13.1 (3.19) | 12.7 (3.12) | 12.6 (3.14) | 12.8 (3.12)
Clinical Global Impressions of Severity (CGI-Severity) score [Mean (Standard Deviation); unit: units on a scale] — CGI-Severity score evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.6 (0.65) | 4.6 (0.65) | 4.6 (0.59) | 4.5 (0.63) | 4.6 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 10 Endpoint
Description: CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. Least Square (LS) means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine 60mg: Duloxetine 60mg orally, once daily for 10 weeks
- Placebo: Placebo capsules identical in appearance, color, taste, and smell to study drug orally, once daily for 10 weeks
Arm/Group | Duloxetine 60mg | Placebo
Number analyzed (Participants) | 105 | 117
units on a scale | -23.9 (1.30) | -21.6 (1.27)
Statistical Analysis 1: Comparison: Duloxetine 60mg vs Placebo; Test type: Superiority or Other; p = 0.193, Mixed Models Analysis

2. Secondary Outcome: Change From Week 10 in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 36 Endpoint
Description: CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 70 | 78 | 80 | 79
units on a scale | -7.8 (1.04) | -7.4 (1.23) | -10.0 (1.17) | -9.0 (1.84)

3. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 10 Endpoint
Description: as for outcome 1
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine 30mg: Duloxetine 30mg orally, once daily for 10 weeks
- Fluoxetine 20mg: Fluoxetine 20mg orally, once daily for 10 weeks
Arm/Group | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 114 | 112 | 117
units on a scale | -24.6 (1.29) | -22.6 (1.27) | -21.6 (1.27)

4. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Subscale Score at Week 10 Endpoint
Description: CDRS-R Subscale scores include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21. Higher score indicates greater severity of disease. LS means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline values.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60mg | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 105 | 114 | 112 | 117
units on a scale
  Mood | -7.1 (0.44) | -7.2 (0.44) | -6.6 (0.43) | -6.4 (0.43)
  Somatic | -7.6 (0.48) | -7.9 (0.48) | -7.1 (0.47) | -6.4 (0.47)
  Subjective | -3.6 (0.26) | -4.0 (0.26) | -3.5 (0.26) | -3.6 (0.26)
  Behavior | -5.8 (0.36) | -5.6 (0.36) | -5.6 (0.35) | -5.4 (0.35)

5. Secondary Outcome: Change From Week 10 in Children's Depression Rating Scale-Revised (CDRS-R) Subscale Score at Week 36 Endpoint
Description: CDRS-R Subscale scores include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21. Higher score indicates greater severity of disease. LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 70 | 78 | 80 | 79
units on a scale
  Mood | -1.9 (0.43) | -1.9 (0.42) | -2.4 (0.44) | -2.3 (0.59)
  Somatic | -2.8 (0.41) | -2.4 (0.52) | -4.0 (0.47) | -3.2 (0.66)
  Subjective | -1.2 (0.25) | -1.3 (0.19) | -1.5 (0.21) | -1.0 (0.32)
  Behavior | -2.1 (0.30) | -1.8 (0.32) | -2.7 (0.28) | -2.4 (0.50)

6. Secondary Outcome: Change From Baseline in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 10 Endpoint
Description: CGI-Severity evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60mg | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 105 | 114 | 112 | 117
units on a scale | -1.5 (0.12) | -1.5 (0.12) | -1.4 (0.11) | -1.4 (0.11)

7. Secondary Outcome: Change From Week 10 in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 36 Endpoint
Description: CGI-Severity evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 69 | 78 | 81 | 79
units on a scale | -1.1 (0.13) | -0.9 (0.16) | -1.3 (0.12) | -1.0 (0.13)

8. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior Baseline Through Week 10
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Treatment Emergent Suicidal Ideation is worsening or new occurrence of events during treatment compared to lead-in baseline (Week -1 to 0).
Time Frame: Baseline through Week 10
Population: Participants with a baseline and at least one post-baseline C-SSRS suicidal ideation or suicidal behavior score and who are at risk for treatment emergent suicidal ideation or behavior.
Measure: Number; unit: participants
Arm/Group | Duloxetine 60mg | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 105 | 115 | 112 | 117
participants
  Suicidal Ideation | 16 | 11 | 13 | 15
  Suicidal Behavior | 0 | 0 | 1 | 1
  Treatment Emergent Suicidal Ideation | 7 | 6 | 9 | 11

9. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior Week 10 Through Week 36
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Treatment Emergent Suicidal Ideation is worsening or new occurrence of events during treatment compared to lead-in baseline (Week 7-10).
Time Frame: Week 10 through Week 36
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 71 | 78 | 80 | 79
participants
  Suicidal Ideation | 6 | 12 | 8 | 8
  Suicidal Behavior | 2 | 3 | 0 | 1
  Treatment Emergent Suicidal Ideation | 5 | 8 | 7 | 6

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hepatic Laboratory Results Any Time Baseline Through Week 10
Description: Total number of participants with any abnormal post-baseline value, based on all values at scheduled and unscheduled visits. Potentially clinically significant hepatic laboratory results at any time are defined as alanine transaminase (ALT) ≥3 x upper limit of normal (ULN), ALT ≥5 x ULN and ALT ≥10 x ULN, as well as ALT ≥3 x ULN and Total Bilirubin ≥2 x ULN.
Time Frame: Baseline through Week 10
Population: Participants with normal ALT value (ALT<1 x ULN) at last non-missing baseline visit and at least one non-missing post-baseline value.
Measure: Number; unit: participants
Arm/Group | Duloxetine 60mg | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 95 | 98 | 102 | 100
participants
  ALT≥3 x ULN | 0 | 0 | 0 | 0
  ALT≥5 x ULN | 0 | 0 | 0 | 0
  ALT≥10 x ULN | 0 | 0 | 0 | 0
  ALT≥3 x ULN and Total Bilirubin≥2 x ULN | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hepatic Laboratory Results Any Time Week 10 Through Week 36
Description: Total number of participants with any abnormal post-baseline value, based on all values at scheduled and unscheduled visits. Potentially clinically significant hepatic laboratory results at any time are defined as ALT ≥3 x ULN, ALT ≥5 x ULN and ALT ≥10 x ULN, as well as ALT≥3 x ULN and Total Bilirubin ≥2 x ULN.
Time Frame: Week 10 through Week 36
Population: Participants with normal ALT value (ALT<1 x ULN) at last non-missing visit before Week 10 and at least one non-missing post-Week 10 value.
Measure: Number; unit: participants
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 69 | 69 | 77 | 73
participants
  ALT≥3 x ULN | 0 | 0 | 0 | 0
  ALT≥5 x ULN | 0 | 0 | 0 | 0
  ALT≥10 x ULN | 0 | 0 | 0 | 0
  ALT≥3 x ULN and Total Bilirubin≥2 x ULN | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Changes in Systolic Blood Pressure (BP), Diastolic BP, Pulse, and Weight Any Time Baseline Through Week 10
Description: PCS increase in systolic and diastolic BP was defined as increase of ≥5 millimeter mercury (mm Hg) from baseline (BL) high value to a value above the 95th percentile at post-BL; PCS increase of pulse was defined as >140 and increase of ≥15 from BL high value for age 7-11 and >120 and increase of ≥15 from BL high value for age 12-17; PCS decrease of pulse was defined as <60 and a decrease of ≥25 from BL low value for age 7-11 and <50 and a decrease of ≥15 from BL low value for age 12-17; PCS decrease of weight was defined as decrease of at least 3.5% from BL low value.
Time Frame: Baseline through Week 10
Population: Participants with normal baseline value and at least one post-baseline value, and who were at risk for the specific PCS criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine 60mg | Duloxetine 30mg | Fluoxetine 20mg | Placebo
Number analyzed (Participants) | 108 | 116 | 117 | 122
percentage of participants
  Diastolic BP Increase (N=93, 100, 99, 110) | 11.8 | 7.0 | 10.1 | 4.5
  Systolic BP Increase (N=88, 95, 93, 98) | 9.1 | 12.6 | 12.9 | 10.2
  Pulse Decrease (N=100, 108, 108, 112) | 0 | 0 | 0 | 0
  Pulse Increase (N=105, 114, 112, 117) | 0 | 0 | 0 | 0
  Weight Decrease (N=105, 114, 112, 117) | 13.3 | 8.8 | 11.6 | 5.1

13. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Changes in Systolic Blood Pressure (BP), Diastolic BP, Pulse, and Weight Any Time Week 10 Through Week 36
Description: PCS increase in systolic and diastolic BP was defined as increase of ≥5 mm Hg from baseline (BL) high value to a value above the 95th percentile at post-BL; PCS increase of pulse was defined as >140 and increase of ≥15 from BL high value for age 7-11 and >120 and increase of ≥15 from BL high value for age 12-17; PCS decrease of pulse was defined as <60 and a decrease of ≥25 from BL low value for age 7-11 and <50 and a decrease of ≥15 from BL low value for age 12-17; PCS decrease of weight was defined as decrease of at least 3.5% from BL low value.
Time Frame: Week 10 through Week 36
Population: Participates with normal value before week 10 and at least one non-missing post-Week 10 value, and who are at risk for the specific PCS criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine 60 mg / Duloxetine 60-120 mg | Duloxetine 30 mg/Duloxetine 60-120 mg | Fluoxetine 20 mg/Fluoxetine 20-40 mg | Placebo/Duloxetine 60-120 mg
Number analyzed (Participants) | 73 | 80 | 84 | 82
percentage of participants
  Diastolic BP Increase (N=55, 65, 64, 69) | 14.5 | 4.6 | 20.3 | 11.6
  Systolic BP Increase (N=53, 62, 57, 57) | 9.4 | 6.5 | 7.0 | 10.5
  Pulse Decrease (N=68, 75, 76, 73) | 0 | 0 | 0 | 0
  Pulse Increase (N=71, 78, 81, 79) | 1.4 | 0 | 0 | 1.3
  Weight Decrease (N=71, 78, 81, 79) | 2.8 | 9.0 | 3.7 | 13.9

ADVERSE EVENTS:
Groups:
- Duloxetine 60 mg - Acute: Duloxetine 60 mg, orally, once daily for 10 weeks
- Duloxetine 30 mg - Acute: Duloxetine 30 mg, orally, once daily for 10 weeks
- Fluoxetine 20 mg - Acute: Fluoxetine 20 mg, orally, once daily for 10 weeks
- Placebo - Acute: Placebo capsules identical in appearance, color, taste, and smell to study drug, orally, once daily for 10 weeks
- Duloxetine 60 mg - Extension; Placebo/Duloxetine - Extension: Duloxetine 60-120 mg , orally, once daily for 6 months
- Duloxetine 30 mg - Extension: Duloxetine 60-120 mg , orally, once daily for 6 months
  One participant who had completed the acute treatment phase and didn't go into the extension phase, was accidentally dispensed the drug at the last visit of the acute treatment phase. Based on intent-to-treat principal, this participant was included in the extension phase analyses for adverse events (AEs; resulting in one more participant being analyzed for AEs than the number of participants who started the extension phase [see Participant Flow section]).
- Fluoxetine 20 mg - Extension: Fluoxetine 20-40 mg, orally, once daily for 6 months
Arm/Group | Duloxetine 60 mg - Acute | Duloxetine 30 mg - Acute | Fluoxetine 20 mg - Acute | Placebo - Acute | Duloxetine 60 mg - Extension | Duloxetine 30 mg - Extension | Fluoxetine 20 mg - Extension | Placebo/Duloxetine - Extension
Serious Adverse Events (participants affected / at risk) | 4/108 | 2/116 | 6/117 | 2/122 | 3/73 | 2/81 | 1/84 | 4/82
Other Adverse Events (participants affected / at risk) | 76/108 | 66/116 | 69/117 | 71/122 | 49/73 | 46/81 | 45/84 | 52/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60 mg - Acute (N=108) | Duloxetine 30 mg - Acute (N=116) | Fluoxetine 20 mg - Acute (N=117) | Placebo - Acute (N=122) | Duloxetine 60 mg - Extension (N=73) | Duloxetine 30 mg - Extension (N=81) | Fluoxetine 20 mg - Extension (N=84) | Placebo/Duloxetine - Extension (N=82)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis of peripheral lymph nodes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60 mg - Acute (N=108) | Duloxetine 30 mg - Acute (N=116) | Fluoxetine 20 mg - Acute (N=117) | Placebo - Acute (N=122) | Duloxetine 60 mg - Extension (N=73) | Duloxetine 30 mg - Extension (N=81) | Fluoxetine 20 mg - Extension (N=84) | Placebo/Duloxetine - Extension (N=82)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 13 (14) | 10 (10) | 10 (10) | 9 (12) | 6 (8) | 6 (7) | 7 (7) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 9 (9) | 3 (3) | 2 (3) | 1 (1) | 5 (7) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (20) | 21 (22) | 11 (12) | 11 (11) | 6 (7) | 13 (14) | 3 (5) | 8 (10)
Vomiting (Gastrointestinal disorders) | 5 (6) | 7 (8) | 2 (2) | 3 (3) | 4 (4) | 10 (13) | 8 (8) | 8 (9)
Fatigue (General disorders) | 5 (5) | 6 (7) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 6 (7)
Pyrexia (General disorders) | 1 (1) | 3 (4) | 0 (0) | 4 (4) | 3 (3) | 3 (4) | 1 (1) | 8 (8)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 7 (8) | 3 (3) | 3 (3) | 6 (7) | 7 (8) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (7) | 3 (3) | 6 (6) | 5 (7) | 4 (6) | 2 (2) | 2 (3)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 5 (5) | 3 (3) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 10 (10) | 6 (6) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 9 (9) | 10 (11) | 5 (5) | 8 (8) | 2 (2) | 6 (6) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 19 (22) | 20 (27) | 22 (26) | 16 (19) | 6 (8) | 4 (4) | 10 (14) | 11 (13)
Somnolence (Nervous system disorders) | 11 (11) | 3 (3) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 6 (6) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days